CLINICAL TRIAL: NCT00063882
Title: A Phase III Study Comparing Combined External Beam Radiation and Transperineal Interstitial Permanent Brachytherapy With Brachytherapy Alone for Selected Patients With Intermediate Risk Prostatic Carcinoma
Brief Title: Interstitial Brachytherapy With or Without External-Beam Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0232; CDR0000288823; NCI-2009-01091 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBRT + Brachytherapy (Experimental): External beam radiation therapy (EBRT) and transperineal interstitial permanent brachytherapy (100/110)
  Interventions: Radiation: Brachytherapy (100/110); Radiation: External Beam Radiation Therapy
- Brachytherapy Only (Active Comparator): Transperineal interstitial permanent brachytherapy (125/145)
  Interventions: Radiation: Brachytherapy (125/145)

INTERVENTIONS:
Radiation: Brachytherapy (100/110) — 100 Gy Palladium-103 (P-102) or 110 Gy Iodine-125 (I-125) seeds within 2-4 weeks of completion of external beam radiotherapy.
  Arms: EBRT + Brachytherapy
Radiation: Brachytherapy (125/145) — 125 Gy Palladium-103 (P-103) or 145 Gy Iodine-125 (I-125) seeds within 4 weeks of study entry.
  Arms: Brachytherapy Only
Radiation: External Beam Radiation Therapy — Total dose of 45 Gy to the prostate and seminal vesicles as a daily dose of 1.8 Gy given 5 times per week. The prescribed dose is defined at the International Commission of Radiation Units and Measurements (ICRU) reference point. Both 3D-conformal radiation therapy (3DCRT) and intensity modulated radiation therapy (IMRT) are permitted.
  Other Names: EBRT
  Arms: EBRT + Brachytherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other sources to damage tumor cells. Interstitial brachytherapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Combining interstitial brachytherapy with external-beam radiation therapy may kill more tumor cells. It is not yet known whether interstitial brachytherapy is more effective with or without external-beam radiation therapy in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of interstitial brachytherapy with or without external-beam radiation therapy in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 5-year freedom from progression in patients with intermediate-risk prostate cancer treated with interstitial brachytherapy with or without external beam radiotherapy (EBRT).
* Compare biochemical (i.e., prostate-specific antigen) failure, biochemical failure by the Phoenix definition, disease-specific survival, local progression, and distant metastases in patients treated with these regimens.
* Compare morbidity and quality of life of patients treated with these regimens.
* Determine the feasibility of collecting Medicare data in a large Radiation Therapy Oncology Group (RTOG) prostate cancer clinical trial for cost effectiveness and cost utility analysis of combined treatment with interstitial brachytherapy and EBRT.
* Prospectively collect diagnostic biopsy samples from these patients for future biomarker analyses.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (T1c vs T2a or T2b), Gleason score (≤ 6 vs 7), prostate-specific antigen (< 10 ng/mL vs 10-20 ng/mL), and prior neoadjuvant hormonal therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo external beam radiotherapy 5 days a week for 5 weeks. Within 2-4 weeks of radiotherapy, patients undergo interstitial brachytherapy with iodine I 125 or palladium Pd 103 seeds.
* Arm II: Patients undergo interstitial brachytherapy only, as in arm I. Quality of life is assessed at baseline, at 4, 12, and 24 months, and then annually for 3 years.

After completion of study treatment, patients are followed at 3-5 weeks, at 4, 6, 9, and 12 months, every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * T1c-T2b, N0, M0
* Intermediate-risk disease, as defined by 1 of the following:

  * Gleason score < 7 AND prostate-specific antigen (PSA) 10-20 ng/mL
  * Gleason score 7 AND PSA < 10 ng/mL
* No evidence of distant metastases
* Prostate volume ≤ 60 cc by transrectal ultrasonography
* American Urological Association voiding symptom score no greater than 15 (alpha blockers allowed)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Patients must use effective contraception
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ at any other site
* No major medical or psychiatric illness that would preclude study therapy
* No hip prosthesis

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Prior neoadjuvant hormonal therapy allowed provided the following are true:

  * Therapy was initiated within 2-6 months of study enrollment
  * Therapy was no more than 6 months in duration
  * Use of 5-alpha reductase inhibitors (e.g., finasteride) is discontinued before registration
* No concurrent hormonal therapy

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* No prior radical surgery for prostate cancer
* No prior transurethral resection of the prostate
* No prior cryosurgery

Other

* No prior transurethral needle ablation of the prostate
* No prior transurethral microwave thermotherapy of the prostate

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2003-06; Primary Completion 2017-05 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley R. Prestidge, MD, Principal Investigator — Bon Secours Cancer Institute
Locations (170):
- United States (168):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente - Division of Research - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Rancho Cordova, Rancho Cordova, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Menorah Medical Center, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Shields Radiation Oncology Center - Mansfield, Mansfield, Massachusetts
  - South Suburban Oncology Center, Quincy, Massachusetts
  - Winchester Hospital Radiation Oncology Center, Winchester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Coleman Radiation Oncology Center at Carter General Hospital, Morehead City, North Carolina
  - CarolinaEast Cancer Care, New Bern, North Carolina
  - South Atlantic Radiation Oncology, LLC, Supply, North Carolina
  - Coastal Carolina Radiation Oncology Center, Wilmington, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Radiation Oncology Center, Alliance, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - St. Francis Hospital, Federal Way, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
- Canada (2):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Michalski JM, Winter KA, Prestidge BR, Sanda MG, Amin M, Bice WS, Gay HA, Ibbott GS, Crook JM, Catton CN, Raben A, Bosch W, Beyer DC, Frank SJ, Papagikos MA, Rosenthal SA, Barthold HJ, Roach M 3rd, Moughan J, Sandler HM. Effect of Brachytherapy With External Beam Radiation Therapy Versus Brachytherapy Alone for Intermediate-Risk Prostate Cancer: NRG Oncology RTOG 0232 Randomized Clinical Trial. J Clin Oncol. 2023 Aug 20;41(24):4035-4044. doi: 10.1200/JCO.22.01856. Epub 2023 Jun 14. PMID 37315297

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Started | 292 | 296
Eligible Patients | 287 | 292
Has Acute Adverse Event Data (Eligible patients who started study treatment) | 282 | 288
Has Late Adverse Event Data (Eligible patients who started study treatment and are alive 181 days after start of radiation) | 282 | 287
Completed (Subjects contributing any data to analysis are considered to have completed the study.) | 287 | 292
Not Completed | 5 | 4
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Eligible Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only | Total
Number analyzed (Participants) | 287 | 292 | 579
Age, Customized [Count of Participants; unit: Participants]
  ≤ 59 | 41 | 51 | 92
  60-69 | 141 | 134 | 275
  70-79 | 102 | 103 | 205
  ≥ 80 | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 287 | 292 | 579
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 274 | 275 | 549
  Unknown or Not Reported | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 5 | 11 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 52 | 102
  White | 223 | 226 | 449
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 1 | 5
Baseline Prostate Specific Antigen (PSA) [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland.
  Participants
    0-<10 ng/ml | 256 | 261 | 517
    10-20 ng/ml | 31 | 31 | 62
Zubrod Performance Status [Count of Participants; unit: Participants] — Measure Description: 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 275 | 281 | 556
    1 | 12 | 11 | 23
Combined Gleason Score (GS) [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    ≤ 6 | 31 | 32 | 63
    7 | 256 | 260 | 516
Gleason Score & PSA [Count of Participants; unit: Participants]
  GS<7 and PSA 10-20 | 31 | 32 | 63
  GS 7 and PSA < 10 | 256 | 260 | 516
T Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1 | 191 | 195 | 386
    T2 | 96 | 97 | 193
Neoadjuvant Hormone Therapy [Count of Participants; unit: Participants]
  Yes | 22 | 25 | 47
  No | 265 | 267 | 532

OUTCOME MEASURES:

1. Primary Outcome: 5-Year Freedom From Progression Rate
Description: A Freedom from Progression (FFP) failure includes biochemical failure, local failure, distant failure, or death due to any cause. Patients who are failure free with less than 5 years of follow-up or who receive any secondary salvage therapy are censored. Freedom from Progression rates are estimated using the Kaplan-Meier method.
Time Frame: From randomization to 5 years
Population: All Eligible Patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
percentage of participants | 85.5 [81.3 to 89.7] | 83.1 [78.7 to 87.5]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Target sample size was 586; 532 patients were needed to test hypothesis of better FFP in the EBRT + Brachytherapy arm over the Brachytherapy Only arm. The trial is designed to detect a 10% improvement in 5-year FFP with 90% power, 1-sided alpha of 0.025. The Z-test statistic for the difference between the 2 5-year FFP rates with the standard errors estimated by Greenwood's method will be used; Test type: Superiority; p = 0.21, Greenwood's T — One-sided significance level of 0.025; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.60 to 1.12] — Reference level = Brachytherapy only

2. Secondary Outcome: Biochemical Failure Rate (Protocol Definition)
Description: Biochemical failure is defined as having 3 consecutive rises of post-treatment PSA or starting hormones after one or more elevations in post-treatment PSA but before 3 consecutive elevations are documented. The sum of the 3 consecutive rises must exceed 1 ng/mL above the nadir. If 3 consecutive PSA rises occur during the first 24 months followed by a subsequent non-hormonal induced PSA decrease, patients will not be considered PSA failures. Three consecutive rises with any of the 3 PSA values occurring more than 24 months after the implant procedure will constitute a failure. Time to biochemical is defined as time from randomization to the date of first biochemical failure, last known follow-up (censored), or death without biochemical failure (competing risk). Biochemical failure rates are estimated using the cumulative incidence method. Five year rates are reported.
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been potentially followed for 5 years. Maximum follow-up at time of analysis was 13.9 years.
Population: All Eligible Patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
percentage of participants | 10.5 [7.2 to 14.4] | 10.5 [7.3 to 14.4]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Test type: Superiority; p = 0.95, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.63 to 1.54] — Reference level = Brachytherapy Only

3. Secondary Outcome: Biochemical Failure (Phoenix Definition)
Description: Biochemical Failure is defined as an increase of 2 ng/ml or more in PSA over the nadir PSA after 24 months from the start of treatment or the start of salvage hormones. Time to biochemical is defined as time from randomization to the date of first biochemical failure, last known follow-up (censored), or death without biochemical failure (competing risk). Biochemical failure rates are estimated using the cumulative incidence method. Five year rates are reported.
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.Maximum follow-up at time of analysis was 13.9 years.
Population: All Eligible Patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
percentage of participants | 8.0 [5.2 to 11.6] | 8.1 [5.3 to 11.7]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Test type: Superiority; p = 0.97, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.64 to 1.58] — Reference level = Brachytherapy Only

4. Secondary Outcome: Prostate Cancer Death
Description: Prostate cancer death is defined as death due to prostate cancer or complications of treatment or death associated with any of the following: 1) further clinical tumor progression occurring after initiation of salvage androgen suppression therapy; 2) a rise that exceeds 1.0 ng/ml in the serum PSA level on at least two consecutive occasions that occurs during or after salvage androgen suppression therapy; and 3) disease progression in the absence of any anti-tumor therapy. Time to prostate cancer death is defined as time from randomization to the date of prostate cancer death, last known follow-up (censored), or death without prostate cancer (competing risk). Prostate cancer death rates are estimated using the cumulative incidence method. Five year rates are reported.
Time Frame: as for outcome 2
Population: All Eligible Patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
percentage of participants | 0.4 [0.0 to 1.9] | 1.1 [0.3 to 2.9]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Test type: Superiority; p = 0.77, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.36 to 3.90] — Reference level = Brachytherapy Only

5. Secondary Outcome: Local Failure
Description: Failure is defined as progression (increase in palpable abnormality) at any time, failure of regression of the palpable tumor by two years, and redevelopment of a palpable abnormality after complete disappearance of previous abnormalities. Histologic criteria for local failure are presence of prostatic carcinoma upon biopsy and positive biopsy of the palpably normal prostate more than two years after the start of treatment. Time to local failure is defined as time from randomization to the date of first local failure, last known follow-up (censored), or death without local failure (competing risk). Local failure rates are estimated using the cumulative incidence method. Five year rates are reported.
Time Frame: as for outcome 2
Population: All Eligible Patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
percentage of participants | 1.5 [0.5 to 3.5] | 1.1 [0.3 to 2.9]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Test type: Superiority; p = 0.99, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.33 to 3.13] — Reference level = Brachytherapy Only

6. Secondary Outcome: Distant Metastases
Description: Failure is defined as the appearance of any distant metastases. Time to distant metastases is defined as time from randomization to the date of first distant metastases, last known follow-up (censored), or death without distant metastases (competing risk). Distant metastases rates are estimated using the cumulative incidence method. Five year rates are reported.
Time Frame: as for outcome 2
Population: All Eligible Patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
percentage of participants | 2.9 [1.4 to 5.4] | 2.1 [0.9 to 4.4]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Test type: Superiority; p = 0.81, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.46 to 2.76] — Reference level = Brachytherapy Only

7. Secondary Outcome: Overall Survival
Description: Failure is defined as death due to any cause. Overall survival time is defined as time from randomization to the date of death or last known follow-up (censored). Survival rates are estimated using the Kaplan-Meier method. Five year rates are reported.
Time Frame: From randomization to last follow-up. Analysis occurs after all patients had been on study for at least 5 years. Maximum follow-up at time of analysis was 13.9 years.
Population: All Eligible Patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
percentage of participants | 95.3 [92.8 to 97.8] | 93.2 [90.3 to 96.2]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Test type: Superiority; p = 0.22, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.51 to 1.17] — Reference level = Brachytherapy Only

8. Secondary Outcome: Percentage of Patients With Acute Grade 2+ and Grade 3+ Toxicities [Genitourinary (GU), Gastrointestinal (GI), and Overall]
Description: Acute toxicities are scored according to NCI Common Toxicity Criteria (CTC) version 2.0 and will be defined as the worst severity of the toxicity occurring ≤ 180 days from start of radiation. The CTC v 2.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to based.
Time Frame: Zero to 180 days from the start of radiation
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 282 | 288
percentage of participants
  Grade 2+ GU/GI | 24.1 [19.5 to 29.4] | 21.9 [17.5 to 27.0]
  Grade 2+ Overall | 27.7 [22.8 to 33.2] | 26.4 [21.6 to 31.8]
  Grade 3+ GU/GI | 6.0 [3.7 to 9.5] | 5.6 [3.4 to 8.9]
  Grade 3+ Overall | 7.8 [5.2 to 11.6] | 8.3 [5.6 to 12.2]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Grade 2+ GU/GI; Test type: Superiority; p = 0.53, Chi-squared — One-sided significance level of 0.05; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.76 to 1.67] — Reference level = Brachytherapy Only
Statistical Analysis 2: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Grade 2+ Overall; Test type: Superiority; p = 0.73, Chi-squared — One-sided significance level of 0.05; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.73 to 1.53] — Reference level = Brachytherapy Only
Statistical Analysis 3: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Grade 3+ GU/GI; Test type: Superiority; p = 0.81, Chi-squared — One-sided significance level of 0.05; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.54 to 2.19] — Reference level = Brachytherapy Only
Statistical Analysis 4: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Grade 3+ Overall; Test type: Superiority; p = 0.82, Chi-squared — One-sided significance level of 0.05; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.51 to 1.69] — Reference level = Brachytherapy Only

9. Secondary Outcome: Time to Late Grade 3+ Toxicities [Genitourinary (GU), Gastrointestinal (GI), and Overall]
Description: Late toxicities are scored according to the Radiation Therapy Oncology Group (RTOG)/European Organisation for Research and Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring Scheme and will be defined as the worst severity of the toxicity occurring > 180 days from radiation start. Grade 3+ GU/GI and overall were analyzed. RTOG/EORTC Late Radiation Morbidity Scoring Scheme assigns Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to toxicity. Time to late grade 3+ toxicity is defined as time from randomization to the date of first late grade 3+ toxicity, last known follow-up (censored), or death without late grade 3+ toxicity (competing risk). Late grade 3+ toxicity rates are estimated using the cumulative incidence method. Five year rates are reported.
Time Frame: From 181 days after the start of radiation to last follow-up. Maximum follow-up at time of analysis was 13.9 years.
Population: Eligible patients who started study treatment and had follow-up data > 180 days from the start of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 282 | 287
percentage of participants
  Grade 3+ GU/GI | 7.9 [5.1 to 11.4] | 3.8 [2.0 to 6.5]
  Grade 3+ Overall | 10.4 [7.2 to 14.3] | 6.6 [4.1 to 9.9]
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Grade 3+ GU/GI; Test type: Superiority; p = 0.01, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 2.37, 95% CI 2-sided [1.20 to 4.68] — Reference level = Brachytherapy Only
Statistical Analysis 2: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Grade 3+ Overall; Test type: Superiority; p = 0.029, Log Rank — One-sided significance level of 0.025; Hazard Ratio (HR) = 1.81, 95% CI 2-sided [1.06 to 3.10] — Reference level = Brachytherapy Only

10. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite (EPIC) From Baseline to 4 Months
Description: The EPIC form is a 50-item, validated tool to assess disease-specific aspects of prostate cancer and its therapies and comprises of four summary domains (bowel, urinary, sexual, and hormonal function). The urinary domain summary score can be separated into 2 distinct subscales: urinary incontinence and urinary irritative. Hormonal domain was excluded as concurrent use of hormones was exclusionary and prior neoadjuvant hormone use was low. Response options for each EPIC item form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life. The change score was calculated as the value at 4 months minus the value at baseline. A negative change reflects a decline at 4 months and a positive change reflects an improvement at 4 months.
Time Frame: Baseline and 4 months after start of radiation
Population: Eligible patients with baseline and 4-month EPIC data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 222 | 241
units on a scale
  Urinary: number analyzed (Participants) | 214 | 234
  Urinary | -20.1 (15.4) | -14.1 (14.8)
  Urinary-Incontinence: number analyzed (Participants) | 204 | 230
  Urinary-Incontinence | -10.3 (17.7) | -8.7 (17.7)
  Urinary-Irritative: number analyzed (Participants) | 211 | 232
  Urinary-Irritative | -23.6 (18.1) | -15.9 (17.3)
  Bowel: number analyzed (Participants) | 218 | 234
  Bowel | -10.4 (13.6) | -6.3 (12.7)
  Sexual: number analyzed (Participants) | 211 | 216
  Sexual | -13.7 (22.3) | -11.2 (21.0)
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Urinary; Test type: Superiority; p < 0.0001, t-test, 2 sided — Significance level of 0.01; Effect size = 0.40 — Minimally important difference (MID) defined as an effect size of at least 0.5. Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7
Statistical Analysis 2: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Urinary- Incontinence; Test type: Superiority; p = 0.33, t-test, 2 sided — significance level of 0.01; Effect size = 0.09 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Urinary-Irritative; Test type: Superiority; p < 0.0001, t-test, 2 sided — significance level of 0.01; Effect size = 0.44 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Bowel; Test type: Superiority; p = 0.001, t-test, 2 sided — significance level of 0.01; Effect size = 0.31 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Sexual; Test type: Superiority; p = 0.23, t-test, 2 sided; Effect size = 0.12; Minimally important difference (MID) defined as an effect size of at least 0.5. Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7

11. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite (EPIC) From Baseline to 24 Months
Description: The EPIC form is a 50-item, validated tool to assess disease-specific aspects of prostate cancer and its therapies and comprises of four summary domains (bowel, urinary, sexual, and hormonal function). The urinary domain summary score can be separated into 2 distinct subscales: urinary incontinence and urinary irritative. Hormonal domain was excluded as concurrent use of hormones was exclusionary and prior neoadjuvant hormone use was low. Response options for each EPIC item form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life. The change score was calculated as the value at 24 months minus the value at baseline. A negative change reflects a decline at 24 months and a positive change reflects an improvement at 24 months.
Time Frame: Baseline and 24 months after start of radiation
Population: Eligible patients with baseline and 24-month EPIC data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 201 | 219
units on a scale
  Urinary: number analyzed (Participants) | 198 | 211
  Urinary | -11.2 (15.7) | -5.6 (13.6)
  Urinary- Incontinence: number analyzed (Participants) | 192 | 207
  Urinary- Incontinence | -7.6 (17.7) | -6.3 (15.5)
  Urinary-Irritative: number analyzed (Participants) | 195 | 210
  Urinary-Irritative | -11.9 (17.4) | -4.8 (14.3)
  Bowel: number analyzed (Participants) | 195 | 213
  Bowel | -7.1 (12.6) | -2.4 (9.9)
  Sexual: number analyzed (Participants) | 190 | 201
  Sexual | -16.7 (23.4) | -10.6 (21.0)
Statistical Analysis 1: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Urinary; Test type: Superiority; p = 0.0002, t-test, 2 sided — Significance level of 0.01; Effect size = 0.38 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Urinary-Incontinence; Test type: Superiority; p = 0.42, t-test, 2 sided — Significance level of 0.01; Effect size = 0.08 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Urinary-Irritative; Test type: Superiority; p < 0.0001, t-test, 2 sided — Significance level of 0.01; Effect size = 0.44 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Bowel; Test type: Superiority; p < 0.0001, t-test, 2 sided — Significance level of 0.01; Effect size = 0.42 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: EBRT + Brachytherapy vs Brachytherapy Only; Sexual; Test type: Superiority; p = 0.0072, t-test, 2 sided — Significance level of 0.01; Effect size = 0.27 — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Change in Total American Urological Association Symptom Index (AUA-SI) Score From Baseline to 4 Months
Description: The AUA-SI is a validated 7-item measure used to assess urinary symptoms. A higher score indicates more severe symptoms for the individual questions and overall total. Six questions ask about frequency of symptoms over the past month with possible responses: 0= Not at all; 1 = Less than 1 time in 5; 2 = less than half the time, 3 = About half the time, 4 = More than half the time, 5 = Almost always. An additional question asks the number of times one gets up to urinate after going to bed, with response indicating the exact number of times ranging from 0 to 5. The total score is the sum of the questions and ranges from 0 to 35. Change is calculated as follow-up timepoint score - baseline score such that a negative change reflects an improvement at the follow-up timepoint and a positive change reflects a decline at the follow-up timepoint.
Time Frame: Baseline and 4 months after start of radiation
Population: Eligible patients who had a total AUA-SI score at baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
units on a scale | 10.12 (7.94) | 7.77 (7.44)

13. Secondary Outcome: Change in Total American Urological Association Symptom Index (AUA-SI) Score From Baseline to 24 Months
Description: as for outcome 12
Time Frame: Baseline and 24 months after start of radiation
Population: Eligible patients who had a total AUA-SI score at baseline and 24 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 223 | 234
units on a scale | 4.54 (6.94) | 2.37 (6.05)

14. Secondary Outcome: Change in European Quality of Life-5 Domains (EQ-5D) From Baseline to 4 Months
Description: The EQ-5D is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 3 problem levels (1-none, 2-moderate, 3-extreme). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm scale ranging from 0 for the worst imaginable health state to 100 for best imaginable health state, marked at 10-point intervals. The change score was calculated as the value at the follow-up timepoint minus the value at baseline. A negative change reflects a decline at the follow-up timepoint and a positive change reflects an improvement at the follow-up timepoint.
Time Frame: Baseline and 4 months after start of radiation
Population: Questionnaires were not completed by all eligible participants. 218 and 227 EBRT + Brachytherapy participants had VAS and index score data, respectively, at baseline and 4 months; 237 and 248 Brachytherapy Only participants had VAS and index score data, respectively, at baseline and 4 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
units on a scale
  VAS Score: number analyzed (Participants) | 218 | 237
  VAS Score | -2.71 (20.26) | -0.44 (17.10)
  Index Score: number analyzed (Participants) | 227 | 248
  Index Score | -0.01 (0.11) | -0.01 (0.12)

15. Secondary Outcome: Change in European Quality of Life-5 Domains (EQ-5D) From Baseline to 24 Months
Description: The EQ5D is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 3 problem levels (1-none, 2-moderate, 3-extreme). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm scale ranging from 0 for the worst imaginable health state to 100 for best imaginable health state, marked at 10-point intervals. The change score was calculated as the value at the follow-up timepoint minus the value at baseline. A negative change reflects a decline at the follow-up timepoint and a positive change reflects an improvement at the follow-up timepoint.
Time Frame: Baseline and 24 months after start of radiation
Population: Questionnaires were not completed by all eligible participants. 210 and 212 EBRT + Brachytherapy participants had VAS and index score data, respectively, at baseline and 24 months; 212 and 226 Brachytherapy Only participants had VAS and index score data, respectively, at baseline and 24 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 287 | 292
units on a scale
  VAS Score: number analyzed (Participants) | 210 | 212
  VAS Score | -0.28 (17.56) | -0.57 (14.94)
  Index Score: number analyzed (Participants) | 212 | 226
  Index Score | -0.02 (0.12) | -0.01 (0.12)

16. Other Pre Specified Outcome: Feasibility of Collecting Medicare Data in a Large RTOG Prostate Cancer Clinical Trial for Cost Effectiveness and Cost Utility Analysis of Combined Treatment With Interstitial Brachytherapy and External Beam Radiotherapy
Time Frame: Analysis occurs after all patients have been potentially followed for 5 years.
Population: The pilot portion of the trial determined that the data required for this analysis was not able to be obtained, and therefore, there are no results for this outcome measure.
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 13.9 years.
Description: Eligible patients who started study treatment are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Groups:
- EBRT + Brachytherapy: 45 Gy EBRT to the prostate and seminal vesicles (1.8 Gy daily over 5 weeks) followed within 2-4 weeks by transperineal interstitial permanent brachytherapy as 100 Gy Palladium-103 (P-102) or 110 Gy Iodine-125 (I-125) seeds.
- Brachytherapy Only: Transperineal interstitial permanent brachytherapy as 125 Gy Palladium-103 (P-103) or 145 Gy Iodine-125 (I-125) seeds within 4 weeks of study entry.
Arm/Group | EBRT + Brachytherapy | Brachytherapy Only
All-Cause Mortality (participants affected / at risk) | 46/282 | 55/288
Serious Adverse Events (participants affected / at risk) | 52/282 | 41/288
Other Adverse Events (participants affected / at risk) | 220/282 | 208/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EBRT + Brachytherapy (N=282) | Brachytherapy Only (N=288)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 | 0
Circulatory or cardiac-Other (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Diarrhea NOS (Gastrointestinal disorders) | 1 | 0
GI-other (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Late RT Toxicity: Other GI : NOS (Gastrointestinal disorders) | 1 | 3
Late RT Toxicity: Small/Large Intestine: NOS (Gastrointestinal disorders) | 6 | 3
Melaena (Gastrointestinal disorders) | 1 | 0
Proctitis NOS (Gastrointestinal disorders) | 0 | 1
Late RT Toxicity: Other : NOS (General disorders) | 14 | 9
Infection NOS (Infections and infestations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Headache NOS (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 2
Late RT Toxicity: Bladder/Other GU : NOS (Renal and urinary disorders) | 22 | 9
Renal/GU-Other (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 10 | 7
Urinary retention (Renal and urinary disorders) | 4 | 4
Impotence (Reproductive system and breast disorders) | 1 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EBRT + Brachytherapy (N=282) | Brachytherapy Only (N=288)
Diarrhea NOS (Gastrointestinal disorders) | 26 | 6
Late RT Toxicity: Other GI : NOS (Gastrointestinal disorders) | 78 | 34
Late RT Toxicity: Small/Large Intestine: NOS (Gastrointestinal disorders) | 88 | 37
Fatigue (General disorders) | 25 | 4
Late RT Toxicity: Other : NOS (General disorders) | 121 | 99
Dysuria (Renal and urinary disorders) | 52 | 28
Late RT Toxicity: Bladder/Other GU : NOS (Renal and urinary disorders) | 160 | 147
Urinary frequency (Renal and urinary disorders) | 96 | 88
Urinary retention (Renal and urinary disorders) | 26 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-12-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT00063882/Prot_SAP_ICF_000.pdf